CLINICAL TRIAL: NCT06102382
Title: The Effect of Two Different Doses of Noradrenaline on Hypotension Caused by Spinal Anesthesia for Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zakaria Ahmed Zakaria, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Noradrenaline in CS under SA
Record Dates: First submitted 2023-10-21; First posted 2023-10-26 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cesarean Section; Hypotension; Norepinephrine
Keywords: Norepinephrine; Spinal anesthesia; Hypotension; Cesarean section
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norepinephrine (0.1) (Experimental): An intravenous bolus dose of norepinephrine (5 µg) followed by infusion of 0.1 µg/kg/min till 5 minutes after delivery of the fetus.
  Interventions: Drug: Norepinephrine (0.1)
- Norepinephrine (0.075) (Active Comparator): An intravenous bolus dose of norepinephrine (5 µg) followed by infusion of 0.075 µg/kg/min till 5 minutes after delivery of the fetus.
  Interventions: Drug: Norepinephrine (0.075)

INTERVENTIONS:
Drug: Norepinephrine (0.1) — An intravenous bolus dose of norepinephrine (5 µg) followed by infusion of 0.1 µg/kg/min till 5 minutes after delivery of the fetus.
  Arms: Norepinephrine (0.1)
Drug: Norepinephrine (0.075) — An intravenous bolus dose of norepinephrine (5 µg) followed by infusion of 0.075 µg/kg/min till 5 minutes after delivery of the fetus.
  Arms: Norepinephrine (0.075)

SUMMARY:
To compare two infusion rates of norepinephrine for prophylaxis against post-spinal hypotension during caesarean delivery.

DETAILED DESCRIPTION:
Hypotension after spinal anesthesia for cesarean delivery is common and is caused mainly by peripheral vasodilatation. Although the intravenous administration of fluids helps, it does not always prevent maternal hypotension. Usually, this hypotension is treated with phenylephrine or ephedrine.

Norepinephrine has been recently introduced for prophylaxis against post-spinal hypotension during cesarean delivery due to its α-adrenergic activity in addition to the weak β-adrenergic activity.

Although the use of norepinephrine for this purpose has shown promising results. However, no sufficient data are available with regard to its optimum dose.

The objective of this study is to compare two infusion rates of norepinephrine for prophylaxis against post-spinal hypotension during caesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women scheduled for cesarean section under spinal anesthesia
* Gestational age of at least 37 weeks

Exclusion Criteria:

* Patient refusal
* Contraindications of spinal anesthesia
* Allergy to the study drug
* Height<150 cm, weight < 60 kg, body mass index (BMI) ≥40 kg/m2.
* patients with cardiac morbidities
* Hypertensive disorders of pregnancy.
* Prepartum hemorrhage

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The frequency of post-spinal hypotension | During the first hour after the subarachnoid block

SECONDARY OUTCOMES:
Arterial blood pressure (Systolic, diastolic, and mean) | During the first hour after the subarachnoid block
Heart rate | During the first hour after the subarachnoid block
Doses of atropine and ephedrine | Intraoperative
Appearance, Pulse, Grimace, Activity, Respiration (APGAR) score | 1, 5, and 10 minutes after delivery
  Ranges from 0 (the worst score) to 10 (the best score)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Woman Health Hospital, Asyut, Egypt